CLINICAL TRIAL: NCT06895993
Title: A Randomized, Open-label, Parallel, Two-treatment, Single Dose Bioequivalence Study of Ferric Carboxymaltose Injection in Healthy Chinese Participants Under Fasting Conditions
Brief Title: Bioequivalence Study of Ferric Carboxymaltose Injection in Healthy Chinese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Huiyu Pharmaceutical Co., Ltd (Industry)
Collaborators: Suzhou Guochen Biotechnology Co., Ltd. (Unknown); Guangzhou Jeeyor Medical Research Co.,Ltd. (Unknown); Boji Medical Technology Co., Ltd. (Unknown); The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024BE-SJMYTT
Record Dates: First submitted 2025-03-20; First posted 2025-03-26 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Healthy Adult
MeSH Terms: interventions — ferric carboxymaltose

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test product-Ferric carboxymaltose Injection provided by SichuanHuiyuPharma (Experimental)
  Interventions: Drug: Ferric Carboxymaltose Injection
- Reference product- licensed by American Regent, Inc. (Active Comparator)
  Interventions: Drug: Ferric Carboxymaltose Injection [Injectafer®]

INTERVENTIONS:
Drug: Ferric Carboxymaltose Injection — For the T group, participants will have a standardized dinner on the night before the trial, followed by a fasting period of at least 10 h before receiving the test product (T, 2 mL: 100 mg elemental iron) via intravenous injection in the single upper limb, at a continuous rate for 1 min, with a speed of 2 mL/min.
  Arms: Test product-Ferric carboxymaltose Injection provided by SichuanHuiyuPharma
Drug: Ferric Carboxymaltose Injection [Injectafer®] — For the R group, participants will have a standardized dinner on the night before the trial, followed by a fasting period of at least 10 h before receiving the reference product (trade name: Injectafer®) (R, 2 mL: 100 mg elemental iron) via intravenous injection on an empty stomach, at a continuous rate for 1 min, with a speed of 2 mL/min.
  Arms: Reference product- licensed by American Regent, Inc.

SUMMARY:
The goal of this clinical trial is to compare the pharmacokinetic profile of the developed drug product and reference product in healthy participants under fasting condition. The main questions it aims to answer are:

* [Question 1] Is there significant difference in the pharmacokinetic profile between the ferric carboxymaltose injection (100 mg iron/2 mL) provided by Sichuan Huiyu Pharmaceutical Co., Ltd. and the ferric carboxymaltose injection licensed by American Regent, Inc. (trade name: Injectafer®, strength: 100 mg iron/2 mL)?
* [Question 2] Is it safe for healthy participants to take ferric carboxymaltose injection (10 mL: 500 mg [calculated by iron]) provided by Sichuan Huiyu Pharmaceutical Co., Ltd. under fasting condition? Participants will be randomly divided into two groups by stratified blocked randomization, with equal number of healthy participants in each group, to receive test product or reference product according to the protocol below.
* Dosing on D1: Group T (Test product) Group R (Reference product)
* PK blood sample collection
* Safety evaluation

ELIGIBILITY:
Inclusion Criteria:

1. Participants must fully understand the purpose, nature, procedures, and potential adverse reactions of the study. They must voluntarily agree to participate in the trial, comply with all study requirements, and provide written informed consent before the initiation of any study procedures.
2. Healthy male or female participants aged 18 to 60 years (inclusive).
3. Male participants must have a body weight of ≥ 50.0 kg. Female participants must have a body weight of ≥ 45.0 kg. BMI must range from 19.0 to 26.0 kg/m² (inclusive).
4. Participants must agree to use highly effective contraceptive measures from screening until 3 months after the last administration. They must have no plans for pregnancy, sperm donation, or egg donation during this period.

Exclusion Criteria:

1. Participants with allergic conditions, such as a known history of hypersensitivity to two or more medications; known allergies to iron, maltose, or its analogues and metabolites; or a history/presence of dermatological conditions (e.g., eczema).
2. History of iron storage diseases (e.g., hemochromatosis), iron utilization disorders (e.g., iron-refractory iron deficiency anemia), hemoglobinopathies (e.g., thalassemia), or symptomatic anemia requiring red blood cell infusion.
3. History of clinically significant acute or chronic, or severe conditions affecting the respiratory, cardiovascular, gastrointestinal, renal, hematological, lymphatic, endocrine, immune, psychiatric, or nervous systems within 12 months prior to screening.
4. Acute infection within 2 weeks prior to screening.
5. Participants with clinically significant abnormalities in vital signs, physical examination, laboratory tests (e.g., hematology, urinalysis, blood chemistry, coagulation function tests, iron metabolism assessments), infectious disease examination, or 12-lead electrocardiogram (ECG), as determined by the investigator; or calcium and phosphorus values in blood chemistry tests are in the abnormal range.
6. Serious arrhythmias shown in ECG at screening, such as recurrent or symptomatic ventricular tachycardia, atrial fibrillation accompanied by rapid ventricular response, or supraventricular tachycardia, and not suitable for the trial at the investigator's discretion.
7. History of hypersensitivity or intolerance to intravenous iron administration.
8. Receiving intravenous iron treatment within 3 months prior to screening, erythropoiesis-stimulating agent (ESA) therapy and/or blood transfusion within 4 weeks prior to screening, and oral iron or iron-containing products within 7 days prior to screening.
9. Use of any medications (prescription, over-the-counter, herbal remedies, or dietary supplements) and healthcare products within 2 weeks prior to screening.
10. History of smoking an average of more than 5 cigarettes per day within 3 months prior to screening or unwillingness to abstain from smoking during the study.
11. Participants who have undergone surgeries within 6 months prior to screening that might affect drug absorption, distribution, metabolism and excretion, or planning to undergo surgeries during the study.
12. Participants who have enrolled in other clinical trials and received investigational products within 3 months prior to screening.
13. Blood donation within 3 months prior to screening; blood donation or significant blood loss due to other reasons within 6 months prior to screening (> 400 mL, excluding menstrual blood loss in female participants), or plan to donate blood during the study.
14. Participants with drug abuse history (including the use of various anesthetic and psychotropic drugs for non-medical purposes) within 1 year prior to screening or have a positive drug abuse test result.
15. Participants with history of alcohol abuse within 1 year prior to screening, defined as average weekly alcohol consume over 2 units (1 unit = 360 mL beer, 45 mL spirits with 40% alcohol, or 150 mL wine), or are unwilling to abstain from alcohol or alcohol-containing products during the study, or have positive breath alcohol test result.
16. Participants who have chocolate, caffeine-containing or xanthine-rich foods or beverages, or specific foods (e.g., animal liver, animal blood, spinach, dragon fruit, mango, grapefruit or grapefruit-containing products), or taking strenuous exercise, or other factors affecting drug absorption, distribution, metabolism, and excretion, within 48 hours before receiving the investigational product.
17. Participants who have received a live vaccine within 14 days prior to screening, or plan to receive vaccination during the study.
18. Inability to tolerate venipuncture or history of fear of needles or hemophobia.
19. Participants with special dietary requirements, and participants who cannot accept the study standardized diet.
20. Participants who have acute illness or receive concomitant medications between screening and investigational product administration.
21. Participants not suitable for the trial at the investigator's discretion.

    In addition to the aforementioned requirements, females who meet the following conditions should also be excluded:
22. Use of oral contraceptives within 30 days prior to screening.
23. Use of long-acting estrogen or progestin injections (progestin-based intrauterine devices), or implants within 6 months prior to screening.
24. Unprotected sexual intercourse with a partner within 14 days prior to screening.
25. Pregnancy, breastfeeding, or positive pregnancy test at screening.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2025-04-07 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2025-05-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter of total iron in serum: Cmax、AUC | 36 hours, 24 hours, and 12 hours before administration; 0 hours and at 5 minutes, 10 minutes, 15 minutes, 30 minutes, 45 minutes, 1 hour, 2 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours, 36 hours, 48 hours, 72 hours, 96 hours post-dose
  Cmax is the peak concentration of total iron in serum. It is directly obtained from observed blood drug concentration-time data. AUC is the area under the concentration curve from dosing to the last measurable blood drug concentration. It is calculated using the linear trapezoidal rule.
Pharmacokinetic parameter of transferrin bound iron in serum: Cmax、AUC | 36 hours, 24 hours, and 12 hours before administration; 0 hours and at 5 minutes, 10 minutes, 15 minutes, 30 minutes, 45 minutes, 1 hour, 2 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours, 36 hours, 48 hours, 72 hours, 96 hours post-dose
  Cmax is the peak concentration of transferrin iron in serum. It is directly obtained from observed blood drug concentration-time data. AUC is the area under the concentration curve from dosing to the last measurable blood drug concentration. It is calculated using the linear trapezoidal rule.

SECONDARY OUTCOMES:
Adverse Events (AEs) and Serious Adverse Events (SAE) | On Day 5
  Safety Assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Phase I clinical trial unit of the First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Undecided